CLINICAL TRIAL: NCT03119623
Title: Prospective Comparison of an ARNI With an ACE Inhibitor on enDOthelial Function by Brachial Artery Reactivity (PARADOR)
Brief Title: Comparing ARNI With ACE Inhibitor on Endothelial Function
Acronym: PARADOR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lost funding prior to study commencing
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Scott David Solomon, Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017P002389/PHS
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; Endothelial function; Brachial Artery Reactivity Test; Sacubitril/Valsartan; Enalapril; HFREF
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril; Enalaprilat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sacubitril/Valsartan (Active Comparator): Sacubitril/valsartan 100mg (Dose Level 1) titrated up if tolerated to 200 mg twice daily (Dose Level 2)
  Interventions: Drug: sacubitril/valsartan
- Enalapril (Active Comparator): Enalapril 5mg (Dose Level 1) titrated up if tolerated to 10mg twice daily (Dose Level 2)
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: sacubitril/valsartan — Sacubitril/valsartan 100mg titrated up to sacubitril/valsartan 200mg
  Other Names: ENTRESTO; LCZ696
  Arms: Sacubitril/Valsartan
Drug: Enalapril — enalapril 5mg, titrated up to 10mg po BID
  Other Names: Vasotec
  Arms: Enalapril

SUMMARY:
PARADOR is multisite, randomized, double-blind, phase IV clinical trial to compare the effect of sacubitril/valsartan (Entresto™) to enalapril (Vasotec®) on blood vessel function in subjects with heart failure with reduced ejection fraction (HFREF).

DETAILED DESCRIPTION:
This multicenter study will enroll 204 adults with a documented diagnosis of heart failure and a documented history of left ventricular ejection fraction.

Subjects will have a screening visit which will last about 2 hours where the following will be done:

* A review of medical history and medications to determine eligibility. An effort will be made to keep doses of other concomitant medication consistent throughout the study.
* Collection of demographic and contact information.
* Vital signs (blood pressure, heart rate, and temperature).
* A urine pregnancy test will be done for women of childbearing potential.
* Blood drawn by venipuncture for safety testing and general health.
* A BART scan of the forearm. The brachial artery vascular reactivity test (BART) is designed to look at the function of the endothelium (the blood vessel lining) using high-resolution ultrasound. This is a non-invasive test. The test is performed with the subject lying down. A blood pressure cuff is placed on the right forearm, just below the bend in the elbow. This cuff is attached to an automatic cuff inflator. The sonographer will hold an ultrasound transducer over the subject's left arm artery (brachial), their upper arm, and measure the size and the blood flow in the artery at baseline. Then the sonographer will inflate a blood pressure cuff over the lower arm for about 5 minutes. After the cuff is released the sonographer will take a picture of the size and blood flow in the artery for 2 minutes after the cuff is released. This test measures the ability of the brachial artery to get bigger (dilate) when exposed to increased blood flow; this ability is a measure of the health of the blood vessel lining. This test may cause temporary numbness and tingling.
* Subjects will be randomized to receive a 2 week supply of enalapril 5mg twice daily or sacubitril/valsartan 49/51 mg twice daily. Subjects will be instructed to take one tablet from each container (active one, one placebo) twice daily. Subjects will be instructed to take their study medication on the day of their BART scan testing.
* If a subject is currently taking an ACE inhibitor, the study team will instruct the subject to HOLD their ACE inhibitor the following day. The subject would then start the study medication at least 36 hours after the missed dose of ACE inhibitor. For example, if study visit is on day 1, subject will HOLD ACE inhibitor morning of day 2, and start taking assigned study medication on study day 3 in the evening. Subjects will continue on their current treatment for their heart condition except for their ACE inhibitor.
* Collection of optional pharmacogenetic blood sample from those subjects agreeing to participate.

Visit 2 (2 week post randomization to study drug), this visit may last 30 minutes where the following will be done:

* A review of medications and changes in medical history.
* Assessment for adverse events and tolerability of study treatment
* Vital signs (blood pressure, heart rate,), if SBP > 105mmHg AND subject is tolerating current study medication dose, titrate to higher study medication dose.
* Collect information regarding changes to concomitant heart failure medications (beta blockers, diuretics, potassium supplement, mineralocorticoid receptor antagonist, other anti-hypertensives). An effort will be made to keep doses of other concomitant medication consistent throughout the study.
* Blood drawn by venipuncture for safety testing.
* Assess study drug adherence (perform a study drug pill count).
* If tolerable, subjects will have their study drugs increased to allow for the target doses of enalpril 10 mg twice daily or sacubitril/valsartan 97/103mg twice daily.
* Dispense 8 weeks of study medication.

Visit 3 (4 week post randomization to study drug), this visit may last 90 minutes where the following will be done:

* A review of medications and changes in medical history.
* Assessment of adverse events and tolerability of study treatment.
* Collect information regarding changes to concomitant heart failure medications (beta blockers, diuretics, potassium supplement, mineralocorticoid receptor antagonist, other anti-hypertensives). An effort will be made to keep doses of other concomitant medication consistent throughout the study.
* Vital signs (blood pressure, heart rate).
* Blood drawn by venipuncture for safety testing.
* Reminded to fast from food, drink, tobacco and to avoid exercise for at least 12 hours prior to Visit 4.

Visit 4 (6 week post randomization to study drug), this visit may last 90 minutes where the following will be done:

* Confirm subject fasted and avoided exercise and tobacco for at least 12 hours.
* A review of medications and changes in medical history.
* Assessment of adverse events and tolerability of study treatment.
* Collect information regarding changes to concomitant heart failure medications (beta blockers, diuretics, potassium supplement, mineralocorticoid receptor antagonist, other anti-hypertensives). An effort will be made to keep doses of other concomitant medication consistent throughout the study.
* Vital signs (blood pressure, heart rate, and temperature).
* A BART scan of the forearm.
* Blood drawn by venipuncture for safety testing.
* Assess study drug adherence (perform a study drug pill count).
* Reminded to fast from food, drink, tobacco and to avoid exercise for at least 12 hours prior to Visit 5.

Visit 5 (10 week post randomization to study drug and end of treatment), this visit may last 90 minutes where the following will be done:

* Confirm subject fasted and avoided exercise and tobacco for at least 12 hours.
* A review of medications and changes in medical history.
* Assessment of adverse events and tolerability of study treatment.
* Collect information regarding changes to concomitant heart failure medications (beta blockers, diuretics, potassium supplement, mineralocorticoid receptor antagonist, other anti-hypertensives). An effort will be made to keep doses of other concomitant medication consistent throughout the study.
* Vital signs (blood pressure, heart rate, and temperature).
* A BART scan of the forearm.
* Blood drawn by venipuncture for safety testing.
* Collect unused study medication.
* Discuss the plan to transition from the study medication to standard of care treatment per the discretion of heart heart failure provider and the subject. Information will be given to the provider and patient regarding results of the PARADIGM-HF trial and updated ACC/AHA/HFSA heart failure treatment guideline update. The study team will instruct the subject to re-start their standard of care ACE inhibitor at least 36 hours after their last dose of study medication. For example, if the subject takes their last dose of study medication on day 70, the subject will wait one day (day 71) and then re-start their standard of care ACE inhibitor day 72 in the evening.
* Schedule visit 6 telephone follow up call

Visit 6 (4 weeks after Visit 5) this visit is a follow-up phone call that may last about 10 minutes where the following will be done:

* A review of medications and changes in medical history.
* Assessment of adverse events.
* Document subject study completion

Early Withdrawal Visit

* Collect study drug.
* Assessment of adverse events
* Collect information regarding changes to concomitant heart failure medications
* Discuss the plan to transition from the study medication to standard of care treatment per the discretion of heart heart failure provider and the subject. The study team will instruct the subject to re-start their standard of care ACE inhibitor at least 36 hours after their last dose of study medication.

Some subjects may have additional visits as they may have to be re-schedule if they had not fasted for 12 hours prior to their study visit or have a fever or due to availability of the BART scan.

Optional Pharmacogenomics Study All subjects enrolled in the study will be invited to donate an optional DNA specimen for pharmacogenomics research. Specimens will be used to achieve the following objectives: 1) predict which subjects are more likely to respond to specific drug therapies; 2) predict which subjects are susceptible to developing adverse side effects; and 3) predict which subjects are likely to progress to more severe disease states.

This will involve the collection of an additional tube of blood (one approximately 10 mL sample) for DNA isolation will be obtained at Visit 1. If, however, the blood sample is not collected during Visit 1, it may be collected at any time (after randomization) during the subject's participation in the study. The collection of the sample will occur after the blood is drawn for safety testing and should not add to much additional (about 5 minutes )time to the study visit. Subjects can still participate in the main study, if they choose not to participate in this optional study.

Subject who participate in the optional pharmacogenomics study can choose whether or not to allow their samples to be banked anonymously when the study ends for future unspecified research. Samples will be banked at the UW-Madison School of Pharmacy until the samples are used up. Subjects can withdraw their permission for banking while the study is active, but the samples will be anonymized at the end of the study for banking and thus cannot be withdrawn a that point.

Data Use and Banking After the research study has been completed and the main results have been published, directly identifiable information will removed and the keys linking codes to subject identity will be destroyed, making data withdrawal impossible. The stored data will not be sent to researchers outside of UW-Madison and will be used for future research about blood vessel function and/or heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, at least 18 years of age
* Documented diagnosis of heart failure
* Documented history of left ventricular ejection fraction < 40% in the 6 months of randomization
* NYHA functional class II or III
* Current treatment with an ACEI at a stable dose of at least enalapril 5 mg twice daily or equivalent for at least 30 days
* Stable heart failure medications (ACEi, +/-beta blocker, +/-mineralocorticoid receptor antagonist) for the past 30 days (with the exception of diuretics) Females of childbearing potential must have a negative urine pregnancy test prior to randomization and agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to randomization, for the duration of study participation, and for 7 days following completion of therapy.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* Documented or self-reported history of hereditary or idiopathic angioedema
* History of acute coronary syndrome, cardiac bypass procedure, stroke, or transient ischemic attack within three months of randomization
* Placement of a biventricular pacemaker device within 6 months of randomization
* History of hypersensitivity or allergy to any of the study drugs or drugs of similar chemical classes
* Current use of sacubitril/valsartan
* Previous intolerance to ACE inhibitors
* Baseline Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m2 per the Modification of Diet in Renal Disease (MDRD) formula
* History of bilateral renal artery stenosis
* History of hepatic dysfunction
* Baseline serum potassium greater than 5.2 mmol/L
* Baseline systolic blood pressure less than 110 mmHg or greater than 180 mmHg
* Enrolled in another clinical trial or has used of any investigational drugs, biologics, or devices within 30 days prior to randomization
* Women who are pregnant or breast-feeding
* Not suitable for study participation due to other reasons at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Vasodilation | At study treatment completion (10 weeks)
  To test the hypothesis that sacubitril/valsartan will improve endothelial function compared to enalapril, evidenced by increased flow mediated vasodilation (FMD) measured by brachial artery reactivity test (BART)

SECONDARY OUTCOMES:
B-type natriuretic peptide | At study treatment completion (10 weeks)
  To test the hypothesis that sacubitril/valsartan will decrease N-terminal pro B-type natriuretic peptide (NT-proBNP) concentrations as compared to enalapril

CONTACTS AND LOCATIONS:
Overall Officials: Orly Vardeny, PharmD, MS, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No